CLINICAL TRIAL: NCT03588585
Title: A Prospective, Randomized Comparison of Tension Versus no Tension With Foley Transcervical Catheters for Pre-induction Cervical Ripening
Brief Title: Tension Versus no Tension With Foley Bulb Induction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hawaii Pacific Health (Other)
Responsible Party: Principal Investigator, Holly Olson, Assistant Professor, Hawaii Pacific Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-077
Record Dates: First submitted 2018-06-22; First posted 2018-07-17 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Induction of Labor Affected Fetus / Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tension (Active Comparator): foley balloon will be placed on tension and taped to thigh at 10 cm. Misoprostil will be placed in posterior vaginal vault.
  Interventions: Procedure: Tension
- No tension (Active Comparator): The foley balloon will be loosely taped without tension to the patient's thigh. Misoprostil will be placed in the posterior vaginal vault.
  Interventions: Procedure: NO TENSION

INTERVENTIONS:
Procedure: Tension — Tension applied to catheter and taped firmly to leg.
  Other Names: misoprostil 25 mcg
  Arms: Tension
Procedure: NO TENSION — Foley balloon will be taped loosely to the leg and not placed on tension. All other care will remain the same
  Other Names: misoprostil 25 mcg
  Arms: No tension

SUMMARY:
To compare the application of tension versus no tension in Foley transcervical catheters for pre-induction cervical ripening.

DETAILED DESCRIPTION:
Patients who are scheduled to undergo labor induction will be offered inclusion in the study which will attempt to determine if placing tension on the foley ballon will shorten the interval between induction initiation and delivery.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparas with singleton live intrauterine pregnancies undergoing labor induction at Kapiolani Medical Center for Women and Children.
* Cephalic presentation
* Intact fetal membranes
* Bishop score less than or equal to 6
* Age greater than or equal to 18 years

Exclusion Criteria:

* Multiparas
* Multiple gestation
* Previous uterine/cervical surgery
* Ruptured fetal membranes
* Fetal malpresentation
* Any contraindication to vaginal delivery at time of admission

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2018-04-16 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Time to Delivery | Will measure length of time from beginning of induction with the foley balloon until delivery
  Reduction in time to delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Kapiolani Medical Center for Women and Children, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264